CLINICAL TRIAL: NCT06303427
Title: Effects of Modified Constraint-induced Movement Therapy With and Without Electrical Stimulation on Range of Motion, Muscle Strength, and Motor Function in ERB's Palsy
Brief Title: Effects of Modified Constraint-induced Movement Therapy With and Without Electrical Stimulation in Erb's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0292
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Erb's Palsy
Keywords: Erb's Palsy; Erb Paralysis; Electric Stimulation; Active movement scale; Randomized clinical trial; Motor function
MeSH Terms: conditions — Brachial Plexus Neuropathies | interventions — Electric Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study would be single-blinded as the assessor of the study would be kept blind to the treatment groups to which patients will be allocated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: (Modified constraint-induced movement therapy + electrical stimulation) (Experimental): Group A will include 17 participants. The participants in this group will receive a 60-minute session daily. Each participant will perform 96 sessions (6 times per week over 16 weeks) for 60 minutes daily.
  1. Electrical stimulation for 20 minutes
  2. Routine physical therapy for 10 minutes
  3. Modified constraint-induced movement therapy for 30 minutes.
  Interventions: Other: Modified constraint-induced movement therapy; Other: Electrical stimulation
- Group B: (Modified constraint-induced movement therapy) (Experimental): 17 participants will be included in this group. The participants in this group will also receive a 60-minute session daily (6 times per week over 19 weeks).
  1. Routine physical therapy for 10 minutes.
  2. Modified constraint-induced movement therapy for 50 minutes.
  Interventions: Other: Modified constraint-induced movement therapy

INTERVENTIONS:
Other: Modified constraint-induced movement therapy — The unaffected arm will be restricted by using an upper extremity sling that will strap to the child's trunk with a distal end fastened to prevent the movement of the unaffected limb.
  The modified constraint-induced movement therapy will include these exercises.
  1. Playing with ball.
  2. Playing with modeling clay.
  3. Playing with LEGOS (building towers or different shapes from the toy bricks).
  4. Tearing a paper towel from a roll.
  5. Holding and eating biscuits.
  6. Eating with a spoon.
  7. Drinking from a glass.
  8. Combing hair.
  9. Brushing teeth.
  10. Making bubbles using a bubble blower.
  11. Pulling a toy.
  12. Placing a hat or piece of cloth on the head.
  13. Applying lotion to the trained caregiver.
Other: Electrical stimulation — The participants in this group will first receive a 20-minute session of electrical stimulation (on time of 10 s, off time of 30 s, pulse rate of 35 Hz, the pulse width of 300 µs).
  Arms: Group A: (Modified constraint-induced movement therapy + electrical stimulation)

SUMMARY:
ERB's palsy is an injury of upper section of the brachial plexus (C5-6) leading to an internally rotated and adducted shoulder and a pronated forearm. Modified constraint-induced movement therapy improves the functionality of the affected limb, while electrical stimulation helps in the improvement of active range of motion and muscle strength in ERB's palsy patients. This study aims to investigate the effects of modified constraint-induced movement therapy with and without electrical stimulation on range of motion, muscle strength, and motor functions in patients with ERB's Palsy.

DETAILED DESCRIPTION:
This randomized clinical trial will be conducted at the Children's Hospital. The sample size will consist of 34 participants. Participants who meet the inclusion criteria will be randomly allocated into two groups using an online randomization tool; Group A will receive modified constraint-induced movement therapy with electrical stimulation and Group B will receive modified constraint-induced movement therapy only. Both groups will receive routine physical therapy as a part of treatment. All participants will receive a 60-minute session, 6 times a week for 16 weeks.

Universal Goniometer will be used to assess range of motion, the Medical Research Council Scale for muscle strength, and the Active Movement Scale for motor function at baseline, 4th, 8th, 12th, and 16th weeks after treatment discontinuation. The data will be analyzed using SPSS version 26 for Windows software.

ELIGIBILITY:
Inclusion Criteria:

1. Children with a confirmed diagnosis of ERB's palsy.
2. Muscle power of the affected limb should be between 1 to 4.
3. Active finger range of motion,10-degree wrist extension, and thumb abduction.

Exclusion Criteria:

1. Children having contracture and stiffness of affected limb.
2. Muscle power of affected limb 0 or 5.
3. Children with cerebral palsy, visual, hearing, and cognitive problems, or any neuromuscular, and skeletal disorders.
4. Previous history of neurological and orthopedic surgery

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Standard universal goniometer | 16 weeks
  It is a device used to measure the range of motion of joints. It consists of four parts: body, fulcrum, stationary, and the moving arm.
Medical Research Council (MRC) Scale | 16 weeks
  It is scale used for testing muscle strength, ranging from Grade 5 (movement through full ROM with maximum resistance against gravity), Grade 4 (movement through full ROM with moderate resistance against gravity), Grade 3 (movement through full ROM without resistance against gravity), Grade 2 (movement through full ROM with gravity eliminated), Grade 1 (flicker of movement) to Grade 0 (no apparent contraction).
Active Movement Scale | 16 weeks
  It is used to quantify movement and assess upper limb motor function. It assesses 15 joint motions (range of motion and muscle strength) from the shoulder to the hand on an 8-point scale (0 ¼ no muscle tone or contraction when gravity is removed, 7 ¼ full range against gravity).

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Kashif, PhD-PT, Study Chair — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zielinski IM, van Delft R, Voorman JM, Geurts ACH, Steenbergen B, Aarts PBM. The effects of modified constraint-induced movement therapy combined with intensive bimanual training in children with brachial plexus birth injury: a retrospective data base study. Disabil Rehabil. 2021 Aug;43(16):2275-2284. doi: 10.1080/09638288.2019.1697381. Epub 2019 Dec 8. PMID 31814455
- [Background] Coroneos CJ, Voineskos SH, Christakis MK, Thoma A, Bain JR, Brouwers MC; Canadian OBPI Working Group. Obstetrical brachial plexus injury (OBPI): Canada's national clinical practice guideline. BMJ Open. 2017 Jan 27;7(1):e014141. doi: 10.1136/bmjopen-2016-014141. PMID 28132014
- [Background] Frade F, Gomez-Salgado J, Jacobsohn L, Florindo-Silva F. Rehabilitation of Neonatal Brachial Plexus Palsy: Integrative Literature Review. J Clin Med. 2019 Jul 5;8(7):980. doi: 10.3390/jcm8070980. PMID 31284431
- [Background] Palomo R, Sanchez R. [Physiotherapy applied to the upper extremity in 0 to 10-year-old children with obstetric brachial palsy: a systematic review]. Rev Neurol. 2020 Jul 1;71(1):1-10. doi: 10.33588/rn.7101.2020029. Spanish. PMID 32583409
- [Background] Sicari M, Longhi M, D'Angelo G, Boetto V, Lavorato A, Cocchini L, Beatrici M, Battiston B, Garbossa D, Massazza G, Titolo P. Modified constraint induced movement therapy in children with obstetric brachial plexus palsy: a systematic review. Eur J Phys Rehabil Med. 2022 Feb;58(1):43-50. doi: 10.23736/S1973-9087.21.06886-6. Epub 2021 Nov 8. PMID 34747579
- [Background] Chang KW, Justice D, Chung KC, Yang LJ. A systematic review of evaluation methods for neonatal brachial plexus palsy: a review. J Neurosurg Pediatr. 2013 Oct;12(4):395-405. doi: 10.3171/2013.6.PEDS12630. Epub 2013 Aug 9. PMID 23930602
- [Background] Van der Looven R, Le Roy L, Tanghe E, Samijn B, Roets E, Pauwels N, Deschepper E, De Muynck M, Vingerhoets G, Van den Broeck C. Risk factors for neonatal brachial plexus palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2020 Jun;62(6):673-683. doi: 10.1111/dmcn.14381. Epub 2019 Oct 31. PMID 31670385
- [Background] de Matos MA, Souto DO, Soares BA, de Oliveira VC, Leite HR, Camargos ACR. Effectiveness of Physical Therapy Interventions in Children with Brachial Plexus Birth Injury: A Systematic Review. Dev Neurorehabil. 2023 Jan;26(1):52-62. doi: 10.1080/17518423.2022.2099995. Epub 2022 Jul 17. PMID 35848401
- [Background] Lewis SP, Sweeney JK. Comorbidities in Infants and Children with Neonatal Brachial Plexus Palsy: A Scoping Review to Inform Multisystem Screening. Phys Occup Ther Pediatr. 2023;43(5):503-527. doi: 10.1080/01942638.2023.2169091. Epub 2023 Jan 19. PMID 36659827
- [Background] Eren B, Karadag Saygi E, Tokgoz D, Akdeniz Leblebicier M. Modified constraint-induced movement therapy during hospitalization in children with perinatal brachial plexus palsy: A randomized controlled trial. J Hand Ther. 2020 Jul-Sep;33(3):418-425. doi: 10.1016/j.jht.2019.12.008. Epub 2020 Mar 7. PMID 32151503
- [Background] Brady K, Garcia T. Constraint-induced movement therapy (CIMT): pediatric applications. Dev Disabil Res Rev. 2009;15(2):102-11. doi: 10.1002/ddrr.59. PMID 19489088